CLINICAL TRIAL: NCT04398108
Title: An Open-Label, Single-arm, Phase I Study to Evaluate the Pharmacokinetics, Tolerability and Safety of Margetuximab Plus Chemotherapy in the Treatment of Chinese Patients With HER2+ Metastatic Breast Cancer Who Have Received Prior Anti-HER2 Therapies
Brief Title: A Study to Evaluate the Pharmacokinetics of Margetuximab in Chinese Patients With HER2+ MBC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zai Lab (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Zai Lab (Hong Kong), Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZL-MG-BC-001
Record Dates: First submitted 2020-05-08; First posted 2020-05-21 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: HER2 Positive Metastatic Breast Cancer
Keywords: Metastatic Breast Cancer; MBC; HER2; Margetuximab
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Margetuximab & Chosen Chemotherapy (Experimental): The dosage and administering of margetuximab is 15 mg/kg IV every 21 days. Investigators need to choose one of the 3 chemotherapies based on patient conditions.
  Interventions: Drug: Margetuximab Margetuximab-IV

INTERVENTIONS:
Drug: Margetuximab Margetuximab-IV — Drug: Chosen Chemotherapy (Capecitabine) -Oral Capecitabine tablet Drug: Chosen Chemotherapy (Vinorelbine) Vinorelbine -IV Drug: Chosen Chemotherapy (Gemcitabine) Gemcitabine -IV

SUMMARY:
This is an open-label, Single-arm, Phase I clinical study to evaluate the pharmacokinetics, tolerability and safety of margetuximab plus chemotherapy in Chinese patients with advanced HER2+ breast cancer who have received standard anti-HER2 directed therapy in the metastatic setting (mandatory including trastuzumab).

The primary endpoint of this study is PK parameters of margetuximab.

DETAILED DESCRIPTION:
Approximately 16~20 Chinese subjects will be enrolled. Eligible subjects are HER2 positive, metastatic breast cancer who has received standard anti-HER2 directed therapy in the metastatic setting in Chinese patients. Subjects should have received treatment with at least one, and no more than four lines of therapy overall in the metastatic setting.

Eligible subjects will receive margetuximab plus chemotherapy. The dosage and administering of margetuximab is 15 mg/kg IV Q3W. Investigators selected one of three backbone chemotherapy regimens given at standard doses: capecitabine, vinorelbine or gemcitabine. Subject will receive the treatment until disease progression, unacceptable toxicity, withdrawal of consent, initiation of subsequent anti-tumor treatment therapy, or death (whichever occurs first).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained prior to performing any protocol-related procedures
* Male or female, age ≥ 18 years old at the time of screening.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Subject has histologically confirmed HER2 positive metastatic breast cancer.
* Have received standard anti-HER2 directed therapy in the metastatic setting (mandatory to have trastuzumab), regardless of having received (neo)adjuvant anti-HER2 therapy or not.
* Have received treatment with no more than four lines of therapy overall in the metastatic setting (including anti-HER2 targeted therapy or chemotherapy) and must have disease progressed on or after, the most recent line of therapy. per RECIST 1.1.
* Previous adverse events associated with anti-tumor therapy have been recovered to NCI-CTCAE v4.03 Grade ≤1 (except NCI-CTCAE v4.03 Grade ≤2 alopecia, stable sensory neuropathy, or stabilized electrolyte disturbance after fluid transfusion).
* Subject has life expectancy ≥12 weeks.
* Subject has no supportive therapy of blood transfusion or growth factor within 4 weeks before dosed and has adequate organ functions
* Subject has a negative test result of pregnancy test at screening.

Exclusion Criteria:

* Subject has symptomatic, uncontrolled brain or pia mater metastasis.
* Subject has third interstitial effusion that cannot be controlled by drainage or other means.
* Subject has local or systemic anti-tumor treatment within 2 weeks prior to enrollment
* Subject has any investigational treatment within 4 weeks prior to enrollment (including margetuximab)
* Subject has history of major surgery with unrecovered surgical effect within 4 weeks prior to enrollment
* Subject has other malignant tumor (complete cured in situ cervical cancer, cutaneous basal cell carcinoma or cutaneous squamous cell carcinoma are not included) within 5 years prior to enrollment
* Subject has severe and uncontrolled disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-08-25 (Actual); Primary Completion 2021-04-27 (Actual); Study Completion 2021-04-27 (Actual)

PRIMARY OUTCOMES:
Evaluation of pharmacokinetic parameter of margetuximab Cmax | Approximately 18 months after the first subject is randomized; anticipated evaluation Jul 2020
Evaluation of pharmacokinetic parameter of margetuximab Tmax | Approximately 18 months after the first subject is randomized; anticipated evaluation Jul 2020
Evaluation of pharmacokinetic parameter of margetuximab T1/2 | Approximately 18 months after the first subject is randomized; anticipated evaluation Jul 2020
Evaluation of pharmacokinetic parameter of margetuximab AUC | Approximately 18 months after the first subject is randomized; anticipated evaluation Jul 2020

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Approximately 18 months after the first subject is randomized; anticipated evaluation Jul 2020
  Incidence of Treatment-Emergent Adverse Events as assessed by CTC AE 4.03

CONTACTS AND LOCATIONS:
Overall Officials: Zeifei Jiang, Principal Investigator — The fifth medical center of the General Hospital of people's Liberation Army of China; Min Yan, Principal Investigator — Henan Cancer Hospital; Cuizhi Geng, Principal Investigator — Hebei Medical University Fourth Hospital
Locations (3):
- China (3):
  - The fifth medical center of the General Hospital of people's Liberation Army of China, Beijing, Beijing Municipality
  - The fourth hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Henan Cancer Hospital, Zhengzhou, Henan